CLINICAL TRIAL: NCT06765967
Title: The Effect of Virtual Reality and Music Recital on Anxiety and Agitation in Patients Undergoing Spinal Anaesthesia: A Randomised Controlled Study
Brief Title: The Effect of Virtual Reality and Music Recital on Anxiety and Agitation in Patients Undergoing Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Semra ERDAĞI ORAL, associate professor doctor, Kafkas University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAFKASSERDAGIORAL-001
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Spinal Anaesthesia; Anxiety State; Surgery; Ajitation
Keywords: spinal anaesthesia; anxiety; patient
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality glasses (Experimental): Patients were shown walking in the forest, underwater life, nature landscapes and snow landscapes with virtual reality goggles.
  Interventions: Other: displaying virtual reality images
- music (Experimental): Music was played to the patients with headphones.
  Interventions: Other: music playback
- control (No Intervention): Patients in the normal operation process, no intervention was performed.

INTERVENTIONS:
Other: displaying virtual reality images — Patients were shown content filmed in 4K resolution through the glasses.
  Other Names: VR
  Arms: virtual reality glasses
Other: music playback — With the permission of the Turkish Music Research and Promotion Group (TÜMATA), 'Acemaşiran Makamı' was played.
  Arms: music

SUMMARY:
This study will be carried out in patients undergoing spinal anaesthesia. The effects of virtual reality and music playback on anxiety and agitation in patients will be evaluated.

DETAILED DESCRIPTION:
Virtual reality is a computer technology in which a virtual environment is simulated in three dimensions. This technology isolates the individual from real life by zooming the lenses to the patient's eyes through a headset known as virtual reality glasses. Recently, with technological developments, virtual reality applications have started to take place among nursing practices as non-pharmacological approaches that support pharmacological methods in clinical settings. Various studies have revealed that virtual reality as a distraction method plays an important role in alleviating anxiety and agitation experienced by patients.

Music application is an easy-to-apply and non-invasive non-pharmacological method. Music recitals give a feeling of relaxation by increasing the release of endorphin hormone in individuals and play an important role as a psychosocial intervention. Such activities reduce symptoms of anxiety and depression, improve quality of life and have positive effects on physical symptoms and general well-being. In addition, the effects of music on respiratory rate, blood pressure and heart rate are also observed.

This study aims to evaluate the effects of virtual reality technology and music playback on anxiety, agitation and physiological parameters in patients undergoing spinal anaesthesia and to make important contributions to the literature in this context.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Clear consciousness, able to communicate,
* No hearing-speech problems,
* Who volunteered to participate in the study,
* Patients who would undergo Urology, General Surgery, Orthopedics, Cardiovascular Surgery, Neurosurgery by spinal anaesthesia were included in the study.

Exclusion Criteria:

* Patients without spinal anaesthesia,
* Patients who participated in the study but voluntarily withdrew at any stage of the study or patients who had to withdraw involuntarily during the operation were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Spinal Anaesthesia Anxiety and Agitation Scale | 1 year
  to evaluate anxiety and agitation in individuals under spinal anaesthesia. Spinal Anaesthesia Anxiety Scale consists of two sub-dimensions called 'Intellectual Experience' and 'Sensory Experience' and 14 questions. The Sensory Experience sub-dimension includes eight questions and the Intellectual Experience sub-dimension includes six questions. The Spinal Anaesthesia Anxiety Scale is a 5-point Likert-type scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree). Spinal Anaesthesia Agitation Scale consisted of 9 questions and three sub-dimensions as 'Verbal Non-Aggressive Behaviours', 'Aggressive Behaviours towards Personnel' and 'Aggressive Behaviours towards Self'.

CONTACTS AND LOCATIONS:
Locations (1):
- Kars Harakani State Hospital Operating Theatre Unit, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No